CLINICAL TRIAL: NCT06158451
Title: Clinical and Radiographic Evaluation of Zinc Oxide-Propolis Mixture Versus Modified Triple Antibiotic Paste in Lesion Sterilization and Tissue Repair (LSTR) for the Treatment of Necrotic Primary Molars: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Zinc Oxide-Propolis Mixture Versus Modified Triple Antibiotic Paste in LSTR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Khaled Adam, Assistant lecturer pediatric dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 208877371
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative; Periapical; Infection
Keywords: propolis; modified triple antibiotic paste; lesion sterilization and tissue repair
MeSH Terms: conditions — Pain, Postoperative; Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc-oxide Propolis (Zno-P) (Experimental): Propolis liquid (Brazilian Green Bee Propolis Liquid Extract, Uniflora®) and Zinc oxide powder will be mixed and added after minimal instrumentation until size 20 to remove all the accessible necrotic pulp and placed on the pulpal floor and intracanal.
  Interventions: Combination Product: Zinc oxide propolis
- Modified triple antibiotic paste (Active Comparator): Metronidazole tablets 500 mg (Flagyl®, Sanofi, Egypt), ciprofloxacin tablets 500 mg (Ciprofloxacin tablets USP 39®, European pharmaceuticals, Egypt,), and clindamycin capsules 300 mg(Dalacin C™ Pfizer, Egypt) will be mixed and added after minimal instrumentation until size 20 to remove all the accessible necrotic pulp and placed on the pulpal floor and intracanal.
  Interventions: Combination Product: Modified triple antibiotic paste

INTERVENTIONS:
Combination Product: Zinc oxide propolis — Propolis liquid (Brazilian Green Bee Propolis Liquid Extract, Uniflora®) and Zinc oxide powder will be mixed on a glass slab with the help of a stainless -steel spatula.
  • The mixing ratio of zinc oxide powder and Propolis liquid is 2:1 until a paste like consistency is reached.
  Arms: Zinc-oxide Propolis (Zno-P)
Combination Product: Modified triple antibiotic paste — Chemotherapeutic agents used are metronidazole tablets 500 mg (Flagyl®, Sanofi, Egypt), ciprofloxacin tablets 500 mg (Ciprofloxacin tablets USP 39®, European pharmaceuticals, Egypt,), and clindamycin capsules 300 mg(Dalacin C™ Pfizer, Egypt).
  * After the removal of enteric coating of tablets with the help of blade, the drugs are pulverized into fine powder using sterilized mortar and pestle.
  * The same amount of each powdered drug (1:1:1) is mixed to form m-TAP powder which is mixed with one part of propylene glycol (P) and the same volume of macrogol (M) to form a paste like consistency
  Arms: Modified triple antibiotic paste

SUMMARY:
The aim of this study is to evaluate and compare the clinical effectiveness of zinc oxide-propolis mixture with triple antibiotic paste in LSTR as root canal filling material in necrotic primary molars.

DETAILED DESCRIPTION:
The promising results of propolis as a natural antibiotic in previous in- vivo studies made it interesting to combine propolis to the golden standard zinc oxide eugenol as an intracanal medication in pulp affected primary molars and use this mix as a natural substitute to the modified triple antibiotic paste (m-TAP) and therefore overcoming the antibiotic bacterial resistance, allergy and developmental anomalies that might arise in permanent successor teeth from m-TAP usage.

ELIGIBILITY:
Inclusion Criteria:

* Children:

  1. Cooperative children aged 4 -7 years old.
  2. Systemically healthy.
* Teeth:

Clinical criteria:

1. Necrotic primary mandibular second molar teeth.
2. Spontaneous pain or tenderness to percussion
3. Deep carious lesion with pulp exposure.
4. Presence of chronic apical abscess or sinus tract Tooth should be restorable. (Thakur et al., 2021)

Radiographic criteria:

1. Coronal-radiographic evidence of a deep carious lesions or lesion approximating pulp
2. Radicular discontinuity of lamina dura, furcation involvement less than or equal to half of shortest root in vertical dimension. (Thakur et al., 2021)

Exclusion Criteria:

* Children:

  1. With physical or emotional alteration.
  2. Children with systemic disease.
  3. Previous history of allergy to antibiotics used in the study.
  4. Children that will not attend follow up. • Teeth:

  <!-- -->

  1. Non restorable carious primary molars.
  2. Grade III mobility

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 1 year
  Binary outcome measured with direct questioning to the patient
Tenderness to percussion | 1 year
  (binary outcome measured by percussion test using back of the dental mirror
Swelling / sinus tract | 1 year
  binary outcome measured with visual examination of the patient examination of the patient
Mobility | 1 year
  (measured by mobility test) and according to Miller's Grades; reduction in grade of mobility from preoperative baseline was treated as success

SECONDARY OUTCOMES:
Radiographic success | 6 months
  The amount of furcation / periapical radiolucency in comparison to preoperative remained static or decreased

CONTACTS AND LOCATIONS:
Overall Officials: Sherine Badr, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No
Data may be provided upon request